CLINICAL TRIAL: NCT02887690
Title: Pilot Project to Evaluate the Revolutionizing Prosthetics Modular Prosthetic Limb System for Upper Extremity Amputees
Acronym: MPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Johns Hopkins University (Other); Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 386304
Record Dates: First submitted 2016-08-18; First posted 2016-09-02 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Prosthesis Use; Limb Loss
Keywords: MPL; prosthetic limb; upper extremity; prosthesis

ARMS (1):
- Modular Prosthetic Limb (Experimental): The Defense Advanced Research Projects Agency's (DARPA) advanced upper limb prosthesis, the Modular Prosthetic Limb (MPL)
  Interventions: Device: Modular Prosthetic Limb

INTERVENTIONS:
Device: Modular Prosthetic Limb
  Other Names: MPL

SUMMARY:
The purpose of this study is to optimize the Defense Advanced Research Projects Agency's (DARPA) advanced upper limb prosthesis, the Modular Prosthetic Limb (MPL), by evaluating the performance, usability, and patient acceptance of the MPL in a clinical setting. This study will be a non-randomized limited clinical optimization study. The study will consist of two phases. Up to twenty-four upper extremity amputees will be recruited in order to ensure twelve subjects for participation in the study: 6 trans-humeral amputees and 6 trans-radial amputees. During Phase 1, subjects will be evaluated for their potential to operate the MPL using a virtual limb controlled by signals from surface electromyograms (sEMG). The first six trans-humeral amputee subjects and the first six trans-radial amputee subjects with a demonstrated proficiency controlling the MPL based on analytical performance metrics will enter Phase 2. During Phase 2, each subject will be fitted for the prosthesis with a custom socket. The user will then evaluate the prosthesis during twelve 1- hour or 1 and one half-hour sessions, working with an occupational therapist and research associates and completing both quantitative and qualitative assessments.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects, 18 to 65 years of age with a unilateral or bilateral upper-limb amputation at any time prior to enrollment
* Active duty military, beneficiary, retiree, and civilian non-beneficiaries are all eligible to participate in this minimal risk study.
* If non active duty military, proof of verified, current health insurance in the form of a health insurance card must be provided in person and health plan expiration date not prior to the end of the projected study participation period will be verified.
* No prior history of vertebral disk disease/condition, sciatica or radiculopathy.
* Ability to follow study instructions and likely to complete all required visits for both phases of the study.
* Normal neurological examination with the exception of limb amputation.
* Medically cleared to use a prosthetic device based on residual limb condition and overall health, including participants both with and without prior prosthetic experience.

Exclusion Criteria

* Age less than 18 or greater than 65.
* Presence of mild to severe traumatic brain injury - permanent or temporary impairments of cognitive, physical, and psychosocial functions with an associated diminished or altered state of consciousness - as indicated by neuropsychological screening that is currently performed routinely on patients by the TBI program at WRNMMCB and noted in the subject's medical record.
* Current, known uncontrolled systemic disease.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Subjects with lack of effort as determined by the research team. Subjects will be screened for effort using the Test of Malingering Memory (TOMM), with a score lower than 42/50 serving as exclusionary.
* Significant Axis I or II diagnosis determined by a neurologist or psychiatrist in the 6 months prior to entry into the study.
* Use of a pacemaker, so as to minimize the risk of surface electromyography interference.
* Lack of health insurance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
MPL functionality during clinical use | From beginning to end of clinical testing period, evaluated up to four weeks
  The overall objective of the study is to determine the functionality of the MPL during clinical use in training scenarios simulating activities of daily living, and to assess patient satisfaction of the MPL by individuals with upper extremity amputations. The results will be used to optimize control and features of the MPL based on qualitative and quantitative user driven feedback in a clinical setting.

SECONDARY OUTCOMES:
Optimally controlled degrees of freedom | From beginning to end of clinical testing period, evaluated up to four weeks
  We will functionally assess the number of optimally controlled degrees of freedom by having users perform comparative assessments using their existing prosthesis as a baseline, followed the MPL configured with increasing number of controllable degrees of freedom to accomplish functional activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Pasquina, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No